CLINICAL TRIAL: NCT04421989
Title: Emotion Coaching Skills as an Augmentation to Family Based Treatment for Adolescents With Anorexia Nervosa: A Pilot Study
Brief Title: Parent Emotion Coaching for Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R34MH115897 (NIH); R34MH115897 (NIH)
Record Dates: First submitted 2020-03-12; First posted 2020-06-09 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa
Keywords: family based treatment; expressed emotion; parent coaching; adolescents
MeSH Terms: conditions — Anorexia Nervosa | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Coaching (Experimental): Participants randomized to FBT + EC parent group condition will also receive FBT as part of their standard of care. In addition to FBT, they will receive 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The EC intervention is designed to reduce expressed emotion (e.g., critical comments) and increase parental warmth. The intervention includes emotional awareness and emotion regulation skills for parents, and emotion communication skills for parents to use with their teens undergoing FBT including active listening, emotion support, labeling emotions, and coping with emotions. The structure of EC parent group sessions will begin with review of homework as applicable, a didactic component to teach new skills, followed by role plays between parents in the group and interventionist, and live coaching and feedback from the interventionist.
  Interventions: Behavioral: Emotion Coaching
- Support Group (Active Comparator): Participants randomized to FBT + Support parent group condition will also receive FBT as part of their standard of care. In addition to FBT, they will receive 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The parent support group facilitates parent discussion and support around a variety of topics central to treatment for pediatric AN including: understanding medical co-morbidities, levels of care for treatment, understanding expected body weight, navigating FMLA, and medications. The facilitator introduces each topic weekly and opens up discussion between parents. The facilitator's role is to ensure the group remains on topic and on time.
  Interventions: Other: Support Group

INTERVENTIONS:
Behavioral: Emotion Coaching — Participants randomized to FBT + EC parent group condition will also receive FBT as part of their standard of care. In addition to FBT, they will receive 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The EC intervention is designed to reduce expressed emotion (e.g., critical comments) and increase parental warmth. The intervention includes emotional awareness and emotion regulation skills for parents, and emotion communication skills for parents to use with their teens undergoing FBT including active listening, emotion support, labeling emotions, and coping with emotions. The structure of EC parent group sessions will begin with review of homework as applicable, a didactic component to teach new skills, followed by role plays between parents in the group and interventionist, and live coaching and feedback from the interventionist.
  Arms: Emotion Coaching
Other: Support Group — Participants randomized to FBT + Support Group parent group condition will also receive FBT as part of their standard of care. In addition to FBT, they will receive 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The support group will have a facilitator introduce each topic weekly and parents will discuss. The facilitator's role is to ensure the group remains on topic and on time. Weekly discussion topics include: co-morbid medical diagnoses, understanding levels of care in treatment, taking time off from work, and medications.
  Arms: Support Group

SUMMARY:
Family based treatment (FBT) is the evidence based treatment for pediatric anorexia nervosa (AN), but 50% of adolescents do not respond and the consequences for non-response are dire (e.g., 11.5% mortality rate). Expressed emotion and parental warmth are significant mechanisms of treatment outcome in adolescents with AN, which are not explicitly targeted by FBT. The current proposal is a parent emotion coaching skills group designed to augment FBT in the treatment of pediatric AN by arming high expressed emotion families with the skills necessary to implement FBT and improve treatment outcomes (e.g., weight restoration).

DETAILED DESCRIPTION:
Pediatric anorexia nervosa (AN) affects 400,000 adolescents in the US with devastating consequences including growth delay, bone density loss, bradycardia, and the highest mortality rate of any psychiatric condition (11.5%), with half of all deaths due to suicide. Early intervention in adolescents is life-saving, making pediatric AN treatment an important public health concern. The goal of pediatric AN treatment is to restore the adolescent back to a healthy weight and reverse the dangerous effects of malnutrition. Family based treatment (FBT) is the gold standard of treatment for pediatric AN; however, 50% of patients do not respond. The consequences of treatment non-response are dire, underscoring the importance of improving treatment via augmentations to address non-response. One barrier to treatment response in pediatric AN is expressed emotion (EE), which is defined as a family's response to an ill patient that is characterized by hostility, critical comments, and emotional overinvolvement. Several studies have highlighted that families with high EE undergoing treatment for their adolescent with AN have poorer outcomes, including higher drop-out rates, lack of weight restoration, and less improvement in eating disorder symptoms. Conversely, parental warmth, a facet of EE, is associated with good outcomes in FBT. Recent parenting interventions focused on emotion coaching (EC) to address high EE have demonstrated success as adjuncts to evidence-based treatments in other pediatric populations (e.g., PTSD, ADHD) but have not been applied to pediatric AN. Given the detrimental effects that high EE has on the re-feeding process and the benefits of parental warmth, emotion coaching has the potential to reduce high EE, increase parental warmth, and improve weight restoration in adolescents with AN. The aim of this R34 pilot effectiveness trial is to evaluate the effectiveness of a FBT + EC parent group intervention in families with high EE. In Stage 1 (Feasibility Stage; Year 1), the investigators will conduct preliminary feasibility and acceptability testing of an EC parent group intervention in 6 patients with pediatric AN and their families who exhibit elevated EE. The data from the Feasibility Stage will be used to modify session content to improve treatment delivery and the uptake of EC skills. Once our manual is refined and finalized, the investigators will conduct a randomized controlled clinical trial (Stage 2) of 50 adolescents and their parents to compare FBT+EC parent group (n=25) versus FBT+support (n=25). The FBT+support condition is a general parent support group that is offered as part of standard care in the CCHMC Eating Disorders Program. FBT will be identical in both the treatment and control conditions, with the EC parent group sessions and parent support group sessions occurring separately from the FBT sessions. If the aims of the project are achieved, this study would have a large impact on pediatric AN with the potential to improve weight restoration outcomes by augmenting FBT for families high in EE.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of AN or AAN
* Must be able to read and speak English
* Must have a caregiver participate who spends at least 50% time with participant

Exclusion Criteria

* Major medical conditions affecting metabolism and/or weight
* Current substance abuse
* Moderate-profound intellectual disabilities
* Active psychosis
* Bipolar disorder

Exclusion Criteria:

Insulin dependent diabetes Thyroid disease

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Aarnio-Peterson, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded from the study before assignment to groups if their caregiver did not screen high in expressed emotion on the Five Minute Speech Sample.
Groups:
- Emotion Coaching: Participants (eligible parent/adolescent dyads) randomized to FBT + EC parent group condition received FBT as part of their standard of care. In addition to FBT, parents (alone without adolescents present) received 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The EC intervention is designed to reduce expressed emotion (e.g., critical comments) and increase parental warmth. The intervention includes emotional awareness and emotion regulation skills for parents, and emotion communication skills for parents to use with their teens undergoing FBT including active listening, emotion support, labeling emotions, and coping with emotions. The structure of EC parent group sessions begins with review of homework as applicable, a didactic component to teach new skills, followed by role plays between parents in the group and interventionist, and live coaching and feedback from the interventionist.
- Support Group: Participants (eligible parent/adolescent dyads) randomized to FBT + Support parent group condition received family based treatment (FBT) as part of their standard of care. In addition to FBT, parents only (without the adolescent) received 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The parent support group facilitates parent discussion and support around a variety of topics central to treatment for pediatric AN including: understanding medical co-morbidities, levels of care for treatment, understanding expected body weight, navigating FMLA, and medications. The facilitator introduces each topic weekly and opens up discussion between parents. The facilitator's role is to ensure the group remains on topic and on time.
Period: Overall Study
Arm/Group | Emotion Coaching | Support Group
Started | 22 (22 caregivers and 22 corresponding adolescents) | 19 (19 caregivers and 19 corresponding adolescents)
Completed | 11 (11 caregivers and 11 corresponding adolescents) | 14 (14 caregivers and 14 corresponding adolescents)
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Population: 22 adolescents and their primary caregivers (n = 22) were randomized to the Emotion Coaching group while 19 adolescents and their primary caregivers (n = 19) were randomized to the Support Group.
Groups:
- Emotion Coaching: Participants (eligible parent/adolescent dyads) randomized to FBT + EC parent group condition received family based treatment (FBT) as part of their standard of care. In addition to FBT, parents only (without adolescents present) received 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The EC intervention is designed to reduce expressed emotion (e.g., critical comments) and increase parental warmth. The intervention includes emotional awareness and emotion regulation skills for parents, and emotion communication skills for parents to use with their teens undergoing FBT including active listening, emotion support, labeling emotions, and coping with emotions. The structure of EC parent group sessions begins with review of homework as applicable, a didactic component to teach new skills, followed by role plays between parents in the group and interventionist, and live coaching and feedback from the interventionist.
- Support Group: Participants (eligible parent/adolescent dyads) randomized to FBT + Support parent group condition received family based treatment (FBT) as part of their standard of care. In addition to FBT, parents only (without adolescents present) received 10 additional, weekly, parent group sessions (each session is 60 minutes, 6-8 group members), within a 3-month time frame to account for cancellations. The parent support group facilitates parent discussion and support around a variety of topics central to treatment for pediatric AN including: understanding medical co-morbidities, levels of care for treatment, understanding expected body weight, navigating FMLA, and medications. The facilitator introduces each topic weekly and opens up discussion between parents. The facilitator's role is to ensure the group remains on topic and on time.
- Total: Total of all reporting groups
Arm/Group | Emotion Coaching | Support Group | Total
Number analyzed (Participants) | 44 | 38 | 82
Age, Categorical [Count of Participants; unit: Participants] — Data characterize adolescent participants and their primary caregiver Population: Data characterizes n = 22 adolescents and their primary caregivers (n = 22) in the Emotion Coaching group and n = 19 adolescents and their primary caregivers (n = 19) in the Support group.
  Participants
    Adolescents: number analyzed (Participants) | 22 | 19 | 41
    Adolescents: <=18 years | 22 | 19 | 41
    Adolescents: Between 18 and 65 years | 0 | 0 | 0
    Adolescents: >=65 years | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 22 | 19 | 41
    Caregivers: <=18 years | 0 | 0 | 0
    Caregivers: Between 18 and 65 years | 22 | 19 | 41
    Caregivers: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Data characterize adolescent participants and their primary caregiver Population: 44 participants in the emotion coaching arm (n = 22 adolescents and their caregivers, n = 22).
  38 participants in the support group arm (n = 19 adolescents and their caregivers, n = 19 caregivers)
  years
    Adolescents: number analyzed (Participants) | 22 | 19 | 41
    Adolescents | 15 (1.6) | 14.7 (1.7) | 14.9 (1.6)
    Caregivers: number analyzed (Participants) | 22 | 19 | 41
    Caregivers | 46.4 (6.5) | 46.2 (6.0) | 46.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Data characterize adolescents and their primary caregiver. Population: We analyzed data from n = 22 Emotion coaching adolescents and their caregivers (n = 22) and n = 19 Support group adolescents and their caregivers (n = 19).
  Participants
    Adolescents: number analyzed (Participants) | 22 | 19 | 41
    Adolescents: Female | 20 | 17 | 37
    Adolescents: Male | 2 | 2 | 4
    Caregivers: number analyzed (Participants) | 22 | 19 | 41
    Caregivers: Female | 22 | 18 | 40
    Caregivers: Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data characterize adolescent participants and their primary caregivers Population: 22 adolescents and their primary caregivers (n = 22) were randomized to the Emotion Coaching group while 19 adolescents and their primary caregivers (n = 19) were randomized to the Support Group.
  Participants
    Adolescents: number analyzed (Participants) | 22 | 19 | 41
    Adolescents: Hispanic or Latino | 1 | 0 | 1
    Adolescents: Not Hispanic or Latino | 21 | 19 | 40
    Adolescents: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 22 | 19 | 41
    Caregivers: Hispanic or Latino | 1 | 0 | 1
    Caregivers: Not Hispanic or Latino | 21 | 19 | 40
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data characterize adolescent participants and their primary caregiver Population: 22 adolescents and their primary caregivers (n = 22) were randomized to the Emotion Coaching group while 19 adolescents and their primary caregivers (n = 19) were randomized to the Support Group.
  Participants
    Adolescents: number analyzed (Participants) | 22 | 19 | 41
    Adolescents: American Indian or Alaska Native | 0 | 0 | 0
    Adolescents: Asian | 0 | 0 | 0
    Adolescents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescents: Black or African American | 0 | 0 | 0
    Adolescents: White | 21 | 19 | 40
    Adolescents: More than one race | 1 | 0 | 1
    Adolescents: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 22 | 19 | 41
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 0 | 0 | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 0 | 0 | 0
    Caregivers: White | 22 | 19 | 41
    Caregivers: More than one race | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Data characterize adolescents participants and their primary caregiver.
  participants
    United States | 44 | 38 | 82
Eating Disorder Examination [Mean (Standard Deviation); unit: units on a scale] — Data characterize adolescent participants. The Eating Disorder Examination assesses behavioral features of eating disorders and severity of eating disorders. The Eating Disorder Examination yields 4 subscales: Restraint, Eating Concerns, Weight Concerns, and Shape Concerns which are then averaged to compute the Global Scale score. Data describe Eating Disorder Examination Global Scale scores. Scores range from 0-6 with higher scores indicating behavioral features of eating disorders (e.g., binge eating & purging), and greater eating disorder severity (e.g., greater weight/shape concerns). Population: Only adolescents completed this measure
  units on a scale
    number analyzed (Participants) | 22 | 19 | 41
    (all) | 3.8 (1.7) | 2.7 (1.5) | 3.3 (1.7)
Five Minute Speech Sample [Mean (Standard Deviation); unit: units on a scale] — Scores characterize primary caregiver levels of criticism and warmth only. The range of possible scores on both Criticism and Warmth is 1-9. Higher Criticism scores indicate greater levels of caregiver criticism towards the adolescent (worse outcome). Higher Warmth scores indicated great levels of caregiver warmth towards the adolescent (better outcome). Population: Only caregivers completed this measure
  units on a scale
    Criticism Score: Coders rate caregiver's critical remarks regarding the adolescent.: number analyzed (Participants) | 22 | 19 | 41
    Criticism Score: Coders rate caregiver's critical remarks regarding the adolescent. | 5.36 (2.3) | 5.26 (1.7) | 5.32 (2.0)
    Warmth Score: Coders rate caregiver's positive remarks regarding the adolescent.: number analyzed (Participants) | 22 | 19 | 41
    Warmth Score: Coders rate caregiver's positive remarks regarding the adolescent. | 5.50 (1.7) | 5.95 (1.8) | 5.71 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Criticism
Description: Parent Criticism was assessed by the Five Minute Speech Sample. This is a recorded five-minute unstructured response that the parent gives when prompted to talk about their feelings about their child. Eligible families will be categorized as high expressed emotion using a modified version of the Family Affective Attitudes Rating Scale (FAARS), which was developed to code the Five Minute Speech Sample in families with adolescents. Scores on Criticism range from 1-9 with higher scores reflective of greater parent criticism towards their adolescent (worse outcome).
Time Frame: baseline, 1-month (halfway through the 10-session emotion coaching intervention), post-treatment, and 3-month follow- up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotion Coaching | Support Group
Number analyzed (Participants) | 11 | 14
score on a scale
  1-Month | 5.5 (2.8) | 3.7 (2.1)
  Post-Treatment | 3.7 (2.0) | 4.3 (2.1)
  3 Month Follow-Up | 2.6 (1.6) | 3.1 (2.0)

2. Primary Outcome: Percent Expected Body Weight (%EBW)
Description: Percent Expected Body Weight is the current weight divided by the adolescent's Expected Body Weight based on their premorbid body mass index percentile for age-and-sex (Body Mass Index Percentile; Centers for Disease Control and Prevention, 2000). Expected Body Weights were calculated by research team members to ensure a standardized calculation methodology. One research team member extracted the highest and lowest premorbid Body Mass Index Percentile from each participant's medical chart and calculated the mean premorbid Body Mass Index Percentile, and Percent Expected Body Weight (i.e., current weight divided by Expected Body Weight). A second coder completed the same process for double data coding. Any discrepancies in weights entered or Expected Body Weight calculations were double checked for accuracy and entered. Higher Percent Expected Body Weight corresponds to better outcomes (e.g., 100% = full weight restoration for individuals with anorexia nervosa).
Time Frame: baseline, 1-month, post-treatment, and 3-month follow up
Measure: Mean (Standard Deviation); unit: percentage of expected body weight
Arm/Group | Emotion Coaching | Support Group
Number analyzed (Participants) | 11 | 14
percentage of expected body weight
  1-Month | 95.1 (7.1) | 90.8 (7.8)
  Post-Treatment | 96.6 (6.3) | 92.5 (8.3)
  3 Month Follow-up | 98.0 (5.6) | 92.6 (10.4)

3. Secondary Outcome: Parental Warmth
Description: Parental Warmth was assessed by the Five Minute Speech Sample. This is a recorded five-minute unstructured response that the parent gives when prompted to talk about their feelings about their child. Eligible families will be categorized as high expressed emotion using a modified version of the Family Affective Attitudes Rating Scale (FAARS), which was developed to code the Five Minute Speech Sample in families with adolescents. Scores on Warmth range from 1-9 with higher scores reflective of greater parent warmth towards their adolescent (better outcome).
Time Frame: baseline, 1-month, post-treatment, and 3 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotion Coaching | Support Group
Number analyzed (Participants) | 11 | 14
score on a scale
  1-Month | 7.0 (1.3) | 6.3 (1.8)
  Post-Treatment | 7.8 (0.6) | 5.5 (1.9)
  3 Month Follow-Up | 7.4 (1.7) | 7.5 (1.6)

ADVERSE EVENTS:
Time Frame: Each adolescent participant was in the study for a duration of 6 months (from consent until follow up assessment).
Description: Adverse events were tracked for adolescent participants only. Caregivers were not monitored/assessed for Adverse Events
Arm/Group | Emotion Coaching | Support Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 2/22 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emotion Coaching (N=22) | Support Group (N=19)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) — Patient was admitted to a psychiatric unit due to suicidal ideation (no attempt)
Acute Food Refusal (Psychiatric disorders) | 0 (0) | 1 (1) — Patient was admitted for medical stabilization due to acute food refusal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT04421989/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04421989/ICF_000.pdf